CLINICAL TRIAL: NCT05813340
Title: Vascularized Inter-positional Periosteal Connective-tissue Flap Versus Collagen Membrane in Guided Bone Regeneration in Horizontal Ridge Augmentation in Aesthetic Zone
Brief Title: Vascularized Inter-positional Periosteal Connective-tissue Flap Versus Collagen Membrane in Guided Bone Regeneration
Acronym: VIP-CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Abdel Hady Ismail, Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111111
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Horizontal Ridge Deficiency
Keywords: VIPCTF; GBR; Horizontal ridge augmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vascularized interpositional periosteal connective tissue flap (Experimental): Vascularized inter-positional periosteal connective tissue flap (VIPCTF) may have many advantages over traditional collagen membranes such as; high vascularity, decreased cost (as it may substitute membrane), providing an increase in soft tissue thickness, and reusability.
  Interventions: Procedure: Vascularized inter-positional periosteal connective tissue flap
- collagen membrane (Active Comparator): Collagen membranes are the most commonly used and can inhibit soft tissue growth in bone defects, They achieve better wound healing and bone regeneration.
  Interventions: Procedure: Vascularized inter-positional periosteal connective tissue flap

INTERVENTIONS:
Procedure: Vascularized inter-positional periosteal connective tissue flap — It is a vascularized pedicled flap derived from the hard palate that can be used as a barrier to prevent in growth of soft tissue in guided bone regeneration and to increase soft tissue quantity

SUMMARY:
this study compares 2 techniques in guided bone regeneration for horizontal ridge augmentation in aesthetic zone

DETAILED DESCRIPTION:
Guided bone regeneration is a technique for ridge augmentation using membranes The membrane of GBR is an essential component of treatment as it has some important characteristics manageability, space-making ability, and adequate mechanical, physical properties, and biocompatibility Collagen membranes are the most commonly used and can inhibit soft tissue growth in bone defects and achieve better wound healing and bone regeneration.

on the other hand, a Vascularized inter-positional periosteal connective tissue flap is a flap that has been used as a substitute for the collagen membrane with promising results. Vascularized inter-positional periosteal connective tissue flap (VIPCTF) may have many advantages over traditional collagen membranes such as; high vascularity, decreased cost (as it may substitute membrane), providing an increase in soft tissue thickness, and reusability.

So Evaluation of effect of vascularized interpositional periosteal connective tissue flap on horizontal ridge augmentation grafting of the anterior maxilla in comaprison with the collagen membranes

ELIGIBILITY:
Inclusion Criteria:

* Patients with a horizontal defect in anterior and premolar areas of the maxilla (aesthetic zone).

Exclusion Criteria:

* poor oral hygiene
* radiation therapy of head and neck cancer
* intraoral soft and hard tissue lesions
* Heavy smoking
* Bone pathology

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Amount of bone width gain (horizontal augmentation) | 6 months
  bone width gain is measured in millimeters by Cone beam computed tomography

SECONDARY OUTCOMES:
Percentage of bone formation in the bone biopsy | 6 months
  Area percentage of newly formed bone is measured through histomorphometric analysis

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Ismail, Maters, Principal Investigator — Cairo University
Locations (1):
- Faculty of dentistry Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khajehahmadi, S., & Rahpeyma, A. (2014). Vascularized interpositional periosteal connective tissue flap in implant dentistry. Journal of Dental Implants, 4(1), 29. https://doi.org/10.4103/0974-6781.130952